CLINICAL TRIAL: NCT01125826
Title: Primary Cell Culture of Surgical Glioma Specimens for Invitro Preclinical Studies
Brief Title: Cell Culture of Glioma Specimens for in Vitro Preclinical Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Yu-Hung Kuo, MD, Neurosciences Institute, Albany Medical College
Other Study IDs: 2536
Record Dates: First submitted 2010-05-18; First posted 2010-05-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All subjects will be give permission for specimen storage by signing a separate permission on the informed consent. All specimens will be stored at a tissue bank for an unspecified amount of time.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to culture primary human brain tumor cells with the specific aims of:

1. Develop primary cultures from human brain tumor surgical specimens
2. Determine the genetic and molecular fingerprints of brain tumors that may have prognostic significance
3. Delineate the mechanisms underlying oncogenesis of brain tumors.
4. Perform in vitro assays with brain tumor derived primary cultures to assess the efficacy of novel therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older undergoing surgical resection for glioma

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older undergoing surgical resection for gliomas.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center, Albany, New York, United States